CLINICAL TRIAL: NCT00902018
Title: The Effect of Eltrombopag on Platelet Survival: the Role of the B-cell L Extra Large (BcL-xL) Pathway
Brief Title: Eltrombopag and the Bcl-extra-large (xL) Pathway in Idiopathic Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0809009980
Record Dates: First submitted 2009-05-08; First posted 2009-05-14 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag; romiplostim

STUDY DESIGN:
Intervention Model Description: 10 patients on eltrombopag and 3 were then treated with romiplostim 10 healthy controls
Oversight: Data Monitoring Committee: No

ARMS (3):
- eltrombopag (Experimental): 10 ITP patients were treated with daily oral eltrombopag 75mg for 2 weeks and complete testing was done at weekly intervals 3 times they then were allowed to receive long-term eltrombopag
  Interventions: Drug: Eltrombopag
- romiplostim (Experimental): 3 of the patients who received eltrombopag were also treated with romiplostim 10 micrograms/kg weekly for 2 weeks with the same complete testing done at weekly intervals three times after a washout period > 1 month they then resumed long-term eltrombopag
  Interventions: Drug: Romiplostim
- healthy controls (Sham Comparator): no intervention single blood draw with complete studies
  Interventions: Other: healthy controls

INTERVENTIONS:
Drug: Eltrombopag — The 10 subjects will be treated with eltrombopag 75 mg once daily. Patients will be monitored 3 times, weekly, for the first 2 weeks, and then monitored as clinically indicated as they continue eltrombopag dosing for 3-4 months.
  Other Names: revolade, promacta
  Arms: eltrombopag
Drug: Romiplostim — three of the patients treated with eltrombopag will be treated with weekly romiplostim at a dose of 10 micrograms/kg weekly for 2 weeks with testing at weekly intervals for 3 times
  Other Names: amg531, nplate
  Arms: romiplostim
Other: healthy controls — single blood draw for all measures included in the intervention arms
  Other Names: volunteers not receiving any treatment
  Arms: healthy controls

SUMMARY:
The purpose of this study is to further evaluate the effects that eltrombopag (and romiplostim) have on platelets in subjects with chronic ITP. Eltrombopag is approved by the Food and Drug Administration (FDA) for the treatment of low platelets in patients with chronic ITP. It is being further studied by GlaxoSmithKline (now Novartis) in other conditions associated with low platelets. This research study is being done because eltrombopag has been shown to increase platelet counts in a different way than other therapies for ITP. The investigators want to further study how eltrombopag and romiplostim affect subjects and their platelets to determine how the study drug should best be used in ITP treatment.

DETAILED DESCRIPTION:
The B-cell lymphoma extra large (Bcl-xL/Bak) balance has been identified as an intrinsic mechanism that is critical in determining platelet lifespan (Mason, Cell 2007). There is evidence that Bcl-xL protein expression in megakaryocytes is regulated by Thrombopoietin (TPO) mediated activation of Akt pathways mediated by Jak2 and Stat 5 (possibly by Stat 3 as well). (e.g., Kozuma et. al., Journal of Thrombosis and Haemostasis). Little is known about the Bcl-xL / Bak axis in patients with ITP, or the effect of TPO-R stimulation on platelet survival in patients with ITP. The TPO effect may be a result of stimulation of thrombopoietin-receptor (TPO-R) signalling in megakaryocytes altering the packaging of Bcl-xl into platelets, or be a direct effect of platelet TPO-R stimulation as described above.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed and dated a written informed consent
* Male or female adults (≥18 years) diagnosed with either primary ITP according to the American Society for Hematology or British Committee for Standards in Haematology (ASH/BCSH) guidelines [Blood, 1996; British Journal of Haematology, 2003] for at least three months prior to study entry or with ITP secondary to Evans syndrome, systemic lupus erythematosus (SLE), or Common Variable Immunodeficiency (including hypogammaglobulinemia).
* Subjects must have responded with a platelet count > 30,000/µL to a previous ITP therapy including thrombopoietic agents.
* Platelet count < 30,000/µL
* Female subjects of childbearing potential are practicing an acceptable method of contraception or are completely abstinent from intercourse.

Exclusion Criteria:

* Active infection
* Previously treated with thrombopoietic agents IF either no response at a therapeutic dose (peak platelet count < 50k) OR treatment with the agent within the past 4 weeks
* Currently treated with concomitant ITP medication that has not been stable in dose for at least 2 weeks - only prednisone, azathioprin, and danazol are allowed.
* Female subjects who are nursing or pregnant
* Thrombosis of any kind within past 6 months or on blood thinners because of thrombosis.
* Intravenous Immunoglobulin (IVIG), IV anti-D, bolus corticosteroids or vinca alkaloids within the past week
* Other cytotoxic or immunosuppressive ITP therapy within the past 8 weeks or rituximab within the past 12 weeks
* Active non-dermatologic malignancy defined as presence of known tumor ie. visible by radiography or evident on blood or bone marrow testing OR receiving chemotherapy within past 2 months
* Hemoglobin < 10 gm/dl or white blood cell count < 2,500/ul
* Liver function tests (ALT, Aspartate Aminotransferase (AST), or total bilirubin) > three times upper limit of normal (ULN)
* Creatinine > two times upper limit of normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2015-09-07 (Actual); Study Completion 2015-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B. Bussel, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Result] Mitchell WB, Pinheiro MP, Boulad N, Kaplan D, Edison MN, Psaila B, Karpoff M, White MJ, Josefsson EC, Kile BT, Bussel JB. Effect of thrombopoietin receptor agonists on the apoptotic profile of platelets in patients with chronic immune thrombocytopenia. Am J Hematol. 2014 Dec;89(12):E228-34. doi: 10.1002/ajh.23832. Epub 2014 Sep 2. PMID 25132654
- See also: Related Info — http://onlinelibrary.wiley.com/doi/10.1002/ajh.23832/abstract

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients with persistent or chronic ITP willing to undergo washout period and then multiple visits (7) in 2 weeks period including 3 larger blood draws
Groups:
- Eltrombopag: Promacta (eltrombopag): Subjects will be treated with eltrombopag 75 mg once daily. Patients will be monitored 3 times a week for the first 2 weeks, and then monitored as clinically indicated as they continue eltrombopag dosing for 3-4 months.
  first blood draw before taking eltrombopag
- Eltombopag Then Romiplostim: patients who receive eltrombopag and then are treated with romiplostim (nplate) to ascertain parallelism between the two agents
- Healthy Volunteer: one blood draw only
Period: Overall Study
Arm/Group | Eltrombopag | Eltombopag Then Romiplostim | Healthy Volunteer
Started | 7 | 3 | 10
Completed | 7 | 3 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 10 patients receive eltrombopag and 3 of these go on to receive romiplostim
Groups:
- Eltrombopag Arm: Participants will be treated with eltrombopag 75 mg once daily. Participants will be monitored three times a week for the first two weeks, and then monitored as clinically indicated as they continue eltrombopag dosing for four months.
- Eltrombopag Receiving Romiplostim: Three Participants who had been on eltrombopag in the past will undergo a washout period and will be treated with Romiplostim 10 ug/kg/weekly for 2 weeks. Participants on Romiplostim will be monitored three times a week for two weeks.
- Healthy Volunteers: single blood draw in healthy volunteers (controls)
- Total: Total of all reporting groups
Arm/Group | Eltrombopag Arm | Eltrombopag Receiving Romiplostim | Healthy Volunteers | Total
Number analyzed (Participants) | 7 | 3 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 10 | 15
  >=65 years | 4 | 1 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 8 | 13
  Male | 4 | 1 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients for Whom Eltrombopag Increases the Platelet Count to > 50,000/uL
Description: number of patients in whom Platelet Counts measured on days 8 and 15 after eltrombopag treatment increase to > 50,000/uL counts on other days are just used to be sure the ones on days 8 and 15 are reasonably accurate and representative
Time Frame: platelet counts on days 8 and 15
Population: 0 participants were analyzed in the healthy control arm because healthy controls did not have any blood draws on day 8 and 15 or receive the intervention and hence data was not collected for these participants
Measure: Number; unit: participants
Groups:
- Eltrombopag Then Romiplostim: Three Participants from Eltrombopag arm will undergo second washout period and will be treated with Romiplostim 10 ug/kg/weekly for 2 weeks. Participants on Romiplostim will be monitored three times a week for two weeks exactly like when they received Eltrombopag.
- Healthy Controls: 10 normal volunteers for a single blood draw
Arm/Group | Eltrombopag Arm | Eltrombopag Then Romiplostim | Healthy Controls
Number analyzed (Participants) | 7 | 3 | 0
participants
  pts with platelet counts > 50,000/uL on day 8 | 6 | 3 |
  Pts with platelet counts > 50,000/uL on day 15 | 6 | 3 |

2. Primary Outcome: Number of Patients Who Received Romiplostim and Increased Their Platelet Counts to > 50,000/uL
Description: number of participants in whom platelet counts measured on day 8 and day 15 after treatment(s) with romiplostim 10 micrograms/kg on days 1 and 8
Time Frame: platelet counts on days 8 and 15
Measure: Number; unit: participants
Groups:
- Romiplostim Treated Patients: 3 patients treated with romiplostim 10 micrograms/kg weekly twice with weekly platelet counts on days 1, 8, and 15
Arm/Group | Romiplostim Treated Patients
Number analyzed (Participants) | 3
participants
  plt cts > 50,000/uL on day 8 | 3
  plt cts > 50,000/uL on day 15 | 3

3. Secondary Outcome: How Many Patients Developed SAEs and/or Abnormal Liver Tests to a Level > 2 Times the Upper Limit of Normal
Description: To assess the safety of eltrombopag, in particular the number of patients with serious adverse events and/or abnormal liver tests reaching a level of more than twice the upper limit of normal for the test these outcomes were assessed periodically for liver tests but other SAEs were not systematically assessed but only with complaints or events
Time Frame: on days 8 and 15
Population: 0 participants were analyzed in the healthy controls arm because healthy controls did not have any blood draw on day 8 and 15 or receive the intervention and hence data was not collected for these participants
Measure: Number; unit: participants
Groups:
- Eltrombopag: 10 ITP patients were treated with daily oral eltrombopag 75mg for 2 weeks and testing was done at weekly intervals 3 times they then were allowed to receive long-term eltrombopag
  Eltrombopag: The 10 subjects will be treated with eltrombopag 75 mg once daily. Patients will be monitored 3 times a week for the first 2 weeks, and then monitored as clinically indicated as they continue eltrombopag dosing for 3-4 months.
- Romiplostim: 3 patients, who first received eltrombopag, were treated with romiplostim 10 micrograms/kg weekly for 2 weeks with the same testing done at weekly intervals three times
  Romiplostim: three of the patients treated with eltrombopag will be treated with weekly romiplostim at a dose of 10 micrograms/kg weekly for 2 weeks with testing at weekly intervals for 3 times and blood counts monitored 3 times per week
Arm/Group | Eltrombopag | Romiplostim | Healthy Controls
Number analyzed (Participants) | 10 | 3 | 0
participants
  number of patients with Abnl LFTs on day 8 | 1 | 0 |
  number of patients Abnl LFTs on day 15 | 1 | 0 |
  number of patients with an SAE on day 8 | 0 | 0 |
  number of patients with an SAE on day 15 | 0 | 0 |

4. Other Pre Specified Outcome: Change From Baseline After Eltrombopag Treatment of Platelet Parameters
Description: Samples were drawn weekly for 2 weeks on days 1, 8, and 15 for the treatment arms and day 1 for the healthy control group. Platelet samples were exposed to small molecule Bcl-xL inhibitor, ABT-737 ex-vivo to explore resistance to apoptosis by determining the half maximal inhibitory concentration (IC50) which was measured for each weekly sample drawn. If the half maximal concentration of ABT737 was increased this meant increased resistance to apoptosis.
  The AKT pathway intermediates were measured since these would indicate the mechanism of the platelet resistance to apoptosis so the two sets of measures confirm each other the AIPF is a measure of how many new platelets are made and the large platelets are similar to that
Time Frame: testing on days 8 and 15
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Eltrombopag Then Romiplostim: Three Participants were treated identically as per the eltrombopag arm and, several months later, would undergo a second washout period and were treated with Romiplostim 10 ug/kg/weekly for 2 weeks.
  Participants on Romiplostim will be monitored as were the Eltrombopag participants for 2 weeks.
- Healthy Control Group: 10 Control Participants without thrombocytopenia or any major health issues were enrolled to provide laboratory comparison data to the ITP patients with a single blood draw for platelet counts, IPF, large platelets, IC50 for apoptosis, AKT pathway intermediates.
Arm/Group | Eltrombopag Arm | Eltrombopag Then Romiplostim | Healthy Control Group
Number analyzed (Participants) | 7 | 3 | 0
Participants
  platelet apoptosis increase on day 8 | 7 | 3 |
  platelet apoptosis increase on day 15 | 2 | 0 |
  increase in intracellular AKT intermediates day 8 | 7 | 3 |
  increase in intracellular AKT intermediates day 15 | 0 | 1 |
  increase in A-IPF day 8 | 7 | 3 |
  increase in A-IPF day 15 | 7 | 3 |
  increase in large platelets day 8 | 7 | 3 |
  increase in large platelets day 15 | 7 | 3 |

ADVERSE EVENTS:
Time Frame: data for investigation collected over 2 weeks in all patients: 7 with eltrombopag alone and 3 with eltrombopag first and, then after a washout period, romiplostim later this would be 10 for eltrombopag and 3 for romiplostim additional medication provided as incentive to patients to enter the study there was a single blood draw without incident in the 10 healthy volunteers
Description: patients were asked for concomitant meds and Adverse Events on every visit
Groups:
- Eltrombopag: Ten participants will be treated with eltrombopag 75 mg once daily. Participants will be monitored three times a week for the first two weeks, and then monitored as clinically indicated as they continue eltrombopag dosing for four months.
- Romiplostim: Three Participants who had been on eltrombopag will undergo a washout period and will be treated with Romiplostim 10 ug/kg/weekly for 2 weeks. Participants on Romiplostim will be monitored three times a week for two weeks.
- Healthy Volunteers: single blood draw in healthy controls/volunteers
Arm/Group | Eltrombopag | Romiplostim | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/3 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/3 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/3 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eltrombopag (N=10) | Romiplostim (N=3) | Healthy Volunteers (N=10)
increase in LFTs (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) — increase in ALT/AST

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes